CLINICAL TRIAL: NCT01927900
Title: THE EFFECTS OF HUMAN-MILK-OLIGOSACCHARIDES ON THE FAECAL MICROBIOTA AND ON GASTROINTESTINAL SYMPTOMS IN HEALTHY VOLUNTEERS A PARALLEL, DOUBLE-BLIND, RANDOMISED, PLACEBO-CONTROLLED DOSE FINDING STUDY
Brief Title: The Effects Of HMO On The Faecal Microbiota And On Gastrointestinal Symptoms In Healthy Volunteers
Acronym: HMO-VOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glycom A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HMO1-2013; SJ-345 (Other: The Scientific Ethical Comitee of Regional Zealand)
Record Dates: First submitted 2013-08-13; First posted 2013-08-23 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Gut Microbiota; Gastrointestinal Symptoms
Keywords: Human milk oligosaccharides; Microbiota; Prebiotics
MeSH Terms: interventions — Health Maintenance Organizations; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- HMO1 (Active Comparator): HMO diluted in water
  Interventions: Dietary Supplement: HMO
- Glucose (Placebo Comparator): Glucose diluted in water
  Interventions: Dietary Supplement: Glucose
- HMO2 (Active Comparator): HMO diluted in water
  Interventions: Dietary Supplement: HMO
- HMO3 (Active Comparator): HMO diluted in water
  Interventions: Dietary Supplement: HMO
- HMO4 (Active Comparator): HMO diluted in water
  Interventions: Dietary Supplement: HMO
- HMO5 (Active Comparator): HMO diluted in water
  Interventions: Dietary Supplement: HMO
- HMO6 (Active Comparator): HMO diluted in water
  Interventions: Dietary Supplement: HMO
- HMO7 (Active Comparator): HMO diluted in water
  Interventions: Dietary Supplement: HMO
- HMO8 (Active Comparator): HMO diluted in water
  Interventions: Dietary Supplement: HMO
- HMO9 (Active Comparator): HMO diluted in water
  Interventions: Dietary Supplement: HMO

INTERVENTIONS:
Dietary Supplement: HMO
  Arms: HMO1; HMO2; HMO3; HMO4; HMO5; HMO6; HMO7; HMO8; HMO9
Dietary Supplement: Glucose
  Arms: Glucose

SUMMARY:
The study is a randomised, placebo-controlled, double-blind, parallel, dose-finding study with healthy volunteers. A total of 100 male and female volunteers will be included. The volunteers will be randomized into one of 10 groups, each of 10 participants, consuming either active product in various mixes and doses (9 groups) or placebo product (1 group) for 2 weeks. The 9 groups receiving active product will receive either one of two Human Milk Oligosaccharides (HMOs) alone or in combination at different doses. The primary purpose of the study is establishing the effects of various compositions and doses of HMOs on the faecal flora and on gastrointestinal symptoms in health adults.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Ability and willingness to understand and comply to the study procedures

Exclusion Criteria:

* Participation in a clinical study one month prior to screening visit and throughout the study.
* Abnormal results of the screening laboratory tests clinically relevant for study participation, as judged by the investigator.
* Any gastrointestinal symptom scored >3 on the GSRS during the screening period
* A mean score on the total GSRS >2 (i.e. above the population norm value) during the screening period
* Any gastrointestinal disease(s) that may cause symptoms or may interfere with the trial outcome, as judged by the investigator.
* Other severe disease(s) such as malignancy, diabetes, severe coronary disease, kidney disease or neurological disease, as judged by the investigator.
* Severe psychiatric disease, as judged by the investigator.
* Use of highly dosed probiotic supplements (yoghurt allowed) 3 months prior to the study and throughout the study.
* Consumption of antibiotic drugs 3 months prior to screening and throughout the study.
* Consumption on a regular basis of medication that might interfere with symptom evaluation (as judged by the investigator) 2 weeks prior to screening and throughout the study.
* Pregnant or lactating or wish to become pregnant during the period of the study.
* Lack of suitability for participation in the study for any reason as judged by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in faecal microbiota | Baseline and after 2 weeks of intake
  Change from baseline in microbiota after 2 weeks of intake
Change from baseline in gastrointestinal symptoms measured with the Gastrointestinal Symptom Rating Scale (GSRS) | Baseline and after 2 weeks of intake
  Change from baseline in GSRS after 2 weeks of intake
Plasma concentration of study product | 0, 3, 6, and 9 hours post intake of study product.
  Detectability of study product in plasma at 0, 3, 6 and 9 hours post intake.
Change from baseline in Bristol Stool form (BSF) scale | Baseline and during intake. Registered daily during study period.
  Change from baseline in BSF during intake
Concentration of study product in urine | 0 and 6 hours post intake
  Detectability of study product in urine 6 hours post intake

SECONDARY OUTCOMES:
Change in specific biomarkers in serum | Baseline and after 2 weeks of intake
  Change from baseline in specific biomarkers in serum after two weeks of intake
Number of participants with adverse events | Baseline to end of the 2 weeks of intake
  Registration of adverse events during intake of study product.
Change in clinical chemistry | Baseline and after 2 weeks of intake
  Change from baseline in clinical chemistry after two weeks of intake.
Change in specific biomarkers in faeces | Baseline and after 2 weeks of intake
  Change from baseline in specific biomarkers in faeces after 2 weeks of intake
Change in haematology | At baseline and after 2 weeks of intake
  Change from baseline in haematology after 2 weeks of intake

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bytzer, MD, Principal Investigator — Department of Medicine, Køge Hospital
Locations (1):
- Department of Medicine, Køge Hospital, Køge, Denmark